CLINICAL TRIAL: NCT00037843
Title: Iodine I-131 Iodocholesterol, Its Use in Adrenal Screening
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NUM88-001
Record Dates: First submitted 2002-05-23; First posted 2002-05-24 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Adrenal Gland Diseases; Adrenal Gland Neoplasms
Keywords: adrenal diseases
MeSH Terms: conditions — Adrenal Gland Diseases; Adrenal Gland Neoplasms

INTERVENTIONS:
Drug: I-131 Iodocholesterol

SUMMARY:
This is a clinical research study using I-131 Iodocholesterol which is an experimental radioactive chemical that when injected into the vein, is picked up in the adrenal glands and permits visualization with gamma imaging devices. These images are used in diagnosing a variety of adrenal abnormalities.Prior to the injection of I-131 Iodocholesterol, the patient will receive perchlorate capsules to block any uptake of I-131 by the thyroid gland if this is deemed important. The patient will continue to take these capsules throughout the period of imaging, which may last up to 1 week. The injection of I-131 Iodocholesterol will be given into a vein and the patient will return for images on at least 1 and possibly 2 occasions between 3-7 days after injection. If the case requires it, the patient may also be given a steroid in tablet form, dexamethasone, to take orally prior to and after the injection to suppress normal adrenal function so that the abnormal tissues can be more easily detected.

ELIGIBILITY:
Adults with suspected adrenal disease, such as adrenal adenoma, carcinoma, hyperplasia, or Addison's Disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 1988-12; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald A. Podoloff, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States